CLINICAL TRIAL: NCT02384369
Title: Phase 2a, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Efficacy, Safety, and Pharmacokinetics of Orally Administered SNC-102 in Subjects With Combat-Related Posttraumatic Stress Disorder Concomitantly Treated With Prazosin
Brief Title: Trial of Oral SNC-102 in Subjects With Combat-Related Posttraumatic Stress Disorder
Acronym: PTSD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient
Sponsor: Synchroneuron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNC-102-221 PT
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Post-Traumatic Stress Disorders; Posttraumatic Stress Disorders; Stress Disorders, Post-Traumatic; Post-Traumatic Stress Disorders, Combat-related
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNC-102 sustained release tablet (Experimental): SNC-102 sustained release tablet for oral administration, 1600 mg BID for 8 weeks
  Interventions: Drug: SNC-102 sustained release tablet
- Placebo (Placebo Comparator): Placebo tablet for oral administration, BID for 8 weeks
  Interventions: Drug: SNC-102 sustained release tablet

INTERVENTIONS:
Drug: SNC-102 sustained release tablet — Sustained release oral tablet of SNC-102
  Other Names: SNC-102; SNC102

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of SNC-102 in adult subjects with cPTSD, added to pre-existing treatment that includes prazosin with or without other psychotropic drugs.

Subjects will be treated with SNC-102 tablets or matching placebo on a BID basis for 8 weeks. Subjects will be evaluated for the symptoms of combat-related posttraumatic stress disorder (cPTSD) as measured by the Clinician Administered PTSD Scale (CAPS-5), compared with the response to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of a diagnosis by a Board-Certified psychiatrist of combat-related posttraumatic stress disorder (cPTSD) according to Diagnostic and Statistical Manual (DSM-5) criteria for PTSD and a history linking the symptoms to combat exposure.
* Taking prazosin for treatment of cPTSD for a minimum of 4 weeks, on a stable dose for at least 2 weeks, and expected to remain on that dose for the duration of the study.
* Having sufficient residual symptoms of PTSD while on the current drug regimen that, in the opinion of the Principal Investigator, additional treatment of the disorder is clinically indicated.
* Body mass index of 18-38 kg/m2 inclusive.

Exclusion Criteria:

* Plans to initiate a new psychotropic medication (other than the study drug) during the period of the study.
* Plans to change the dose or discontinue prazosin or a psychotropic medication during the period of the study.
* Diagnosis of epilepsy or treatment with an antiepileptic drug.
* Use of alcohol or cannabis to the extent that, in the view of the Principal Investigator, it raises a significant risk of medication noncompliance, drinking alcohol after midnight on the days of study visits or missed study visits. Any use of non-prescribed opiates, cocaine, or other street drugs other than cannabis in the month prior to study entry.
* Any history of major medical complications of alcohol use including alcoholic hepatitis, cirrhosis of the liver, pancreatitis, alcohol withdrawal seizures, or delirium tremens.
* Patients taking moderate, stable doses of oral opiates for chronic pain may be admitted at the discretion of the Principal Investigator.
* Current use of a drug other than prazosin with significant alpha-adrenergic blocking effects, if associated with symptomatic orthostatic hypotension.
* Current use of cocaine, amphetamine, phencyclidine, or ketamine, documented either by history or by urinary drug screening at Screening and Baseline Visits. Urinary drug screening for ketamine and phencyclidine will conducted off-site by the Study Sponsor if urinary drug screening available at the study site does not include these drugs. Any other drugs identified incidentally on drug screening will warrant exclusion only if the Principal Investigator, in consultation with the Sponsor, judges that their presence could interfere with the objectives of the trial.
* Pregnant or lactating female.
* Women of childbearing potential, unless the subject agrees to use dual contraceptive methods while on study drug and for 1 month afterward, which, in the opinion of the Principal Investigator, are effective and adequate for that subject's circumstances.
* Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that could increase the risk associated with study participation or study drug administration, could interfere with the informed consent process and/or with compliance with the requirements of the study, or could interfere with the interpretation of study results and which, in the Principal Investigator's opinion, would make the subject inappropriate for entry into this study.
* Use of any non-pharmacologic psychiatric somatic treatment within 4 weeks of baseline, or expected during the course of the study. Such treatments include but are not limited to electroconvulsive therapy, transcranial magnetic stimulation, transcranial direct current stimulation, vagus nerve stimulation, light therapy, and acupuncture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms as measured by Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual-5 (CAPS-5) | 8 weeks
  Determine whether SNC-102 at a dose of 1600 mg twice daily (BID), added to pre-existing treatment that includes prazosin, will decrease the symptoms of combat-related posttraumatic stress disorder (cPTSD) as measured by the CAPS-5, compared with the response to placebo.